CLINICAL TRIAL: NCT05839002
Title: Primary Tumor Burden Score: A Novel Staging Parameter Superior to ypT-category for Esophageal Squamous Cell Carcinoma After Neoadjuvant Chemoradiotherapy
Brief Title: Primary Tumor Burden Score:A Novel Staging Parameter for ESCC After nCRT
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xu Huang, Resident Physician, Fudan University
Other Study IDs: CMISG1708
Record Dates: First submitted 2023-03-29; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Neoplasm, Esophagus; Neoplasm, Squamous Cell
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Patients' pathological sections
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Training cohort will be used to find the best calculation and cut-off values for PTBS in ESCC after nCRT.
  Interventions: Procedure: nCRT
- Validation cohort: The study's conclusion will be verified in Zhongshan Hospital Xiamen branch.
  Interventions: Procedure: nCRT

INTERVENTIONS:
Procedure: nCRT — ESCC patients that recieved surgery and nCRT.

SUMMARY:
In this case-only study, the investigators try to define a novel staging parameter, the Primary Tumor Burden Score (PTBS).

DETAILED DESCRIPTION:
In this case-only study, the investigators try to define a novel staging parameter, the Primary Tumor Burden Score (PTBS), which will combine the proportion of residual primary tumor cells and pre-treatment pathological T stage (prepT stage). The investigators will also try to improve ypTNM stage by results of PTBS.

ELIGIBILITY:
Inclusion Criteria:

- Neoadjuvant chemoradiotherapy and surgical resection of esophageal squamous cell carcinoma

Exclusion Criteria:

* Patients receiving neoadjuvant chemoradiotherapy for esophageal squamous cell carcinoma without surgical resection

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ESCC undergoing nCRT at the Department of Thoracic Surgery, Zhongshan Hospital of Fudan University (training cohort), and the Department of Thoracic Surgery, Zhongshan Hospital Xiamen Branch (validation cohort), between January 2010 and February 2019 were reviewed. The inclusion criteria were (I) thoracic ESCC; (II) McKeown or Ivor-Lewis transthoracic approach; (III) locally advanced resectable tumor with cT3-4aNany staging treated with nCRT; (IV) no history of concomitant or prior malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2010-05-21 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Five-year survival of patients | From surgery to the end of follow-up(at least 5 years later)
  The survival of the patients was recorded by follow-up for five years after surgery.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang X, Jiang D, Sun T, Zhou G, Zeng Z, Zhang S, Lin M, Fan H, Jian Z, You R, Liu F, Wu M, Xu W, Tang H, Hou Y, Tan L. Primary Tumour Burden Score: A Novel Staging Parameter for Oesophageal Squamous Cell Carcinoma after Neoadjuvant Chemoradiotherapy. Eur J Cardiothorac Surg. 2025 Sep 2;67(9):ezaf254. doi: 10.1093/ejcts/ezaf254. PMID 40758472